CLINICAL TRIAL: NCT05277597
Title: Effect of a 4-week Post-exercise Sauna Bathing on Targeted Gut Microbiota and Intestinal Barrier Function in Healthy Men: a Randomized Controlled Pilot Trial
Brief Title: Effect of a 4-week Post-exercise Sauna Bathing on Targeted Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: David C. Nieman (Unknown); Tomasz Cisoń (Unknown); Joanna Szurkowska (Unknown); Mirosława Gałęcka (Unknown); Dariusz Sitkowski (Unknown); Zbigniew Szyguła (Unknown)
Responsible Party: Principal Investigator, Joanna Karolkiewicz, prof. AWF dr hab., Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PoznanUPhyEd 25.02.2020
Record Dates: First submitted 2022-02-28; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Healthy Males
Keywords: gut microbiota, exercise, sauna bathing, intestinal barrier
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study used a randomized, parallel group design. The participants were randomly assigned to exercise training (ET) without or with post-exercise sauna treatments (ET+S) by using a permuted blocks of block size 4. design with a computer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group (ET+S ) (Experimental): Participants exercised 60 minutes, 3 times per week, on a bicycle ergometer followed by a 30-minute dry Finish sauna treatment.
  Interventions: Diagnostic Test: The exercise 60 minutes, 3 times per week, on a bicycle ergometer followed by a 30-minute dry Finish sauna treatment.
- The group (ET) (Active Comparator): Participants exercised 60 minutes, 3 times per week
  Interventions: Diagnostic Test: The same exercise training program without the sauna treatments

INTERVENTIONS:
Diagnostic Test: The exercise 60 minutes, 3 times per week, on a bicycle ergometer followed by a 30-minute dry Finish sauna treatment. — Participants in the group ET+S (n=8) exercised 60 minutes, 3 times per week, on a bicycle ergometer followed by a 30-minute dry Finish sauna treatment.Blood and stool samples were collected before and after the 4-week training program.
  Other Names: ET+S
  Arms: The group (ET+S )
Diagnostic Test: The same exercise training program without the sauna treatments — The control group (ET, n=7) engaged in the same exercise training program without the sauna treatments. Blood and stool samples were collected before and after the 4-week training program.
  Other Names: ET
  Arms: The group (ET)

SUMMARY:
Body temperature fluctuations induced by acute exercise bouts may influence the intestinal barrier with related effects on epithelial permeability, immune responses, and release of metabolites produced by the gut microbiota.

DETAILED DESCRIPTION:
Untrained males aged 22±1.5 years were randomly assigned to exercise training (ET) with or without post-exercise sauna treatments (S). Participants in the group ET+S (n=8) exercised 60 minutes, 3 times per week, on a bicycle ergometer followed by a 30-minute dry Finish sauna treatment. The control group (ET, n=7) engaged in the same exercise training program without the sauna treatments. Blood and stool samples were collected before and after the 4-week training program. Blood samples were analysed for the concentration of high-sensitivity C-reactive protein (hsCRP) and complete blood counts. Stool samples were analysed for pH, quantitative and qualitative measures of targeted bacteria and fungi, zonulin, and secretory immunoglobulin A. This study evaluated the effects of post-exercise sauna bathing in young men undergoing endurance training on gut bacteria inflammation and intestinal barrier function. Investigators hypothesized that sauna bathing applied immediately after a physical training session may impact homeostatic control of the gut microbiota and the function of the intestinal barrier.

ELIGIBILITY:
Inclusion Criteria:

* absence of medical contraindications such as epilepsy,addiction to medicines, alcohol and drugs, cancer, blood clotting disorders,
* no infections in the last 4 weeks prior to the study,
* no injuries in the last 4 weeks prior to the study.

Exclusion Criteria:

* the intake of antibiotics, steroids, oral antifungal agents (except for topical antifungals), antiparasitic agents, pre- and/or probiotics,
* history of travel to tropical countries during the last 4 weeks before the study,
* history of adverse responses to sauna bathing.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Change from abundance of Faecalibacterium prausnitzi of the genus Faecalibacterium, Akkermansia muciniphila of the genus Akkermansia, Bifidobacterium spp. of the genus Actinobacteria and Bacteroides spp. of the genus Bacteroidetes at 4 weeks. | baseline and immediately after the intervention
  Bacterial DNA was isolated from stool samples using the QIAamp Fast DNA Stool Mini Kit (QIAGEN, Danish). The anaerobic bacteria were determined by Real-Time PCR with appropriate primers (ThermoFisher Scientific, USA).The results of quantitative bacterial analysis were converted to the decimal logarithm (Log10). The entire Real-Time PCR methodology was developed and validated by the Institute of Microecology in Herborn, Germany
Change from the concentrations of sIgA (marker of mucosal immunity), and zonulin (marker of intestinal permeability) in stool at 4 weeks. | baseline and immediately after the intervention
  Secretory immunoglobulin A concentrations in stool samples were determined with the Secretory IgA test (ImmuChrom GmbH, Heppenheim, Germany). Zonulin concentrations were assessed using the IKD Zonulin ELISA Kit (Immunodiagnostik AG, Bensheim, Germany).
Change from the concentration of high-sensitivity C-reactive protein (hsCRP) at 4 weeks. | baseline and immediately after the intervention
  The concentration of hsCRP was measured by immunoenzymatic assay using a commercially available kit (DRG International Inc., Springfield Township, NJ, USA).

SECONDARY OUTCOMES:
Change from the white blood cell counts (WBC) and subsets at 4 weeks. | baseline and immediately after the intervention
  Blood samples (approx. 2 ml) were taken from the antecubital vein.Complete blood count indices were determined by flow cytometry with a Synergy 2 SIAFRT analyser (Bio Tek, Winooski, VT, USA).
Change feom cardio-respiratory measures at 4 weeks. | baseline and immediately after the intervention
  Peak oxygen uptake (VO2peak) was assessed with MetaMax 3B analyzer (Cortex, Germany) using a graded exercise test (GXT) with a cycloergometer Cyclus2 (Avantronic, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Karolkiewicz, Prof., Principal Investigator — Poznan University of Physical Education
Locations (1):
- Tomasz Cisoń, Nowy Sącz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karolkiewicz J, Nieman DC, Cison T, Szurkowska J, Galecka M, Sitkowski D, Szygula Z. No effects of a 4-week post-exercise sauna bathing on targeted gut microbiota and intestinal barrier function, and hsCRP in healthy men: a pilot randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Jun 16;14(1):107. doi: 10.1186/s13102-022-00497-z. PMID 35710395